CLINICAL TRIAL: NCT06485648
Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Transfusion for the Treatment of Refractory Lupus Nephritis
Brief Title: Mesenchymal Stem Cell Transfusion for the Treatment of Refractory Lupus Nephritis
Acronym: LN
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Professor, Chief physician, Academician of Chinese Academy of Engineering, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-533; 2020YFA0113004 (Other Grant/Funding Number: National Key Research and Development Program of China)
Record Dates: First submitted 2024-06-15; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; Mesenchymal Stem Cells; Randomized Controlled Trial
MeSH Terms: conditions — Lupus Nephritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Normal saline
- Treatment (Experimental)
  Interventions: Biological: Umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Umbilical cord mesenchymal stem cells — Treatment: G(glucocorticoid) + i.v. uc-MSC (1×106 cells/Kg)
  Arms: Treatment
Drug: Normal saline — Control: G(glucocorticoid) + i.v. Normal saline
  Arms: Control

SUMMARY:
Lupus nephritis (LN) is the most common and serious complication of systemic lupus erythematosus (SLE), which can lead to permanent kidney injury and uremia. At present, the combination of glucocorticoids and immunosuppressants is still the first line of clinical treatments. Only about 20%-30% of patients with LN can achieve a complete response. In addition, attainment of clinical remission does not necessarily reflect improvement in the kidney tissues, A substantial proportion of patients who show a clinical response to treatment still have histological findings in their kidney biopsy samples that are consistent with active kidney disease after clinical complete remission. Because of the complexity of refractory lupus nephritis, there is no uniform and effective treatment for them. Mesenchymal stem cells (MSCs) are a class of pluripotent stem cells, that can secrete hundreds of cytokines to participate in immune regulation, anti-inflammatory and anti-fibrosis processes, etc., so they have been actively explored for the treatment of autoimmune diseases which Including systemic lupus erythematosus and lupus nephritis recently. Therefore, MSCs have been considered as a potential therapeutic regimen for the treatment of refractory LN. Several clinical trials have been performed, but the results have been inconsistent and the outcome indicators of treatment were not verified by pathological findings. Therefore, this trial wishes to investigate whether MSCs can improve renal recovery in patients with refractory lupus nephritis and to evaluate the effectiveness of treatment by renal biopsy.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease in which the immune system loses its immune tolerance to endogenous nuclear substances due to unknown reasons. The incidence and prevalence of SLE in different ethnic groups are different, and the overall incidence and prevalence are about 1.4-8.6/100,000 person-years and 13-366.6/100,000 person, respectively. The incidence and prevalence of SLE in China are about 4-10/100,000 person-years and 97.5-100/100,000 person, respectively. Based on this, it is estimated that there are about 1 million patients with SLE in China, which is a major serious chronic disease. Among patients with systemic lupus erythematosus (SLE), the reported lifetime incidence of lupus nephritis (LN) is 20%-60%, depending on the demographics of the population studied. Kidney involvement in SLE has been associated with higher mortality, especially for patients progressing to kidney failure. The ultimate goal of treating LN is to preserve kidney function and reduce the morbidity and mortality associated with chronic kidney disease (CKD) and kidney failure, while minimizing medication-associated toxicities.

At present, the pathogenesis of LN remains unclear. A genome-wide association study (GWAS) conducted by investigators team found that 9 single nucleotide polymorphism loci were associated with the occurrence of LN. The interaction of multiple factors such as gene polymorphism, viral infection, estrogen, ultraviolet light and smoking leads to increased production and decreased clearance of endogenous nuclear substances inside and outside the kidneys in the body, which induce the imbalance of regulation of innate immune system and adaptive immune system, especially the generation of more long-lived plasma cells, resulting in continuous production of autoantibodies in kidney, and they did not respond to standard immunosuppressive therapy. Deposition of antigen-antibody complexes in all parts of the kidneys, which triggers an inflammatory cascade that includes complement activation and aggregation of various immune cells such as T cells, B cells, dendritic cells (DCs), and macrophages. Many of them have pro-inflammatory phenotypes. These factors eventually put the kidneys in a storm of proinflammation.

The clinical manifestations of LN vary from asymptomatic to nephrotic syndrome, acute nephritis syndrome and chronic nephritis syndrome, but the severity of clinical manifestations does not match the actual pathological involvement of the kidneys. The 2024 EULAR Guideline and the 2024 KDIGO guideline recommend the use of kidney biopsy results as the basis for standard diagnosis and treatment of LN. Currently, according to the 2016 revised International Society of Nephrology/Renal Pathology Society (ISN/RPS) classification system, the pathological manifestations of LN are divided into 6 types (I-VI).

Active LN (National Institutes of Health (NIH) activity index≥1 with or without chronicity index) of Class III, IV or III+V, or IV+V are the focus of clinical treatment. The rationale for classifying LN into different classes is based on differences in the prognosis. Patients with proliferative LN (class III/IV) present the worst prognosis without treatment, and the higher rate of refractory response, and patients with class III, IV, or V LN, but not class I or II LN, are at immediate risk of CKD progression and involve irreversible nephron loss that reduces kidneys lifespan. Immunosuppressive therapy is mostly used for the treatment of class III and class IV and combined with or without class V LN, which is divided into two phases: an induction phase with intensive immunosuppression, usually lasting 3-6 months; and a maintenance phase of prolonged, less intensive treatment to prevent renal flares. The recommended standard first-line treatment for these lesions is as follows: initially with glucocorticoids combined with one of the following options: Calcineurin inhibitors (Voclosporin/Tacrolimus/cyclosporine); Mycophenolic acid analogs (MPAA); Cyclophosphamide; Belimumab+MPAA or reduced-dose cyclophosphamide. The maintenance phase of treatment mainly includes reducing prednisone to <5 mg/d, and combined with mycophenolate mofetil. The treatment efficacy indicators include the following: complete response, partial response, and no kidney response. However, the complete response rate of LN is only 20%-30% after receiving six months of standard treatment, which is far from satisfactory. Refractory lupus nephritis indicates an inadequate response to lupus nephritis therapy. At present, there is no clear definition for refractory cases, which is defined in 2024 KDIGO Guidelines as no kidney response within initial first-line standard treatment.

In recent years, in addition to the first-line standard treatment regimen of glucocorticoid combined with immunosuppressants. More and more biological agents are being developed, including Rituximab, Ocrelizumab, Caplacizumab, Belimumab, Abatacept, Anifrolumab, APL-2, BI 655064, BMS-986165, Iscalimab, Obinutuzumab, etc. With the exception of Belimumab and Rituximab were recommended for the treatment of some patients especially those in refractory cases, most of these drugs are being studied in clinical trials. However, the clinical data of the current treatment are too few, the long-term treatment effects of these drugs are not exact, and more new treatment options are urgently needed.

Mesenchymal stem cells (MSCs) are a class of pluripotent stem cells, that are derived from early-developing mesoderm tissues and can be extracted from bone marrow, umbilical cord, umbilical cord blood, embryo, adipose tissue, and other tissues. More and more studies suggest that MSCs can secrete hundreds of cytokines, chemokines, and signaling molecules involved in immune regulation, and anti-inflammatory and anti-fibrosis processes, so they have been actively explored for the treatment of autoimmune diseases in recent years. The immunomodulatory mechanisms of MSCs have been studied using in vitro and in vivo experimental animal models of many autoimmune disorders. Our previous studies have also shown that MSC can effectively alleviate renal lesions in lupus nephritis mice by regulating the kidney region immunity, especially reduce the number of long-lived plasma cells and decrease the level of autoantibodies secreted locally in the kidney tissue.

At present, more than ten clinical trials of stem cell therapy for LN have been registered on the ClinicalTrial website, and among these two trial results have been published. However, the results of the two clinical trials were inconsistent.

Human Umbilical Cord-Mesenchymal Stem Cells (uc-MSCs) were derived from umbilical cord Wharton jelly, which are non-invasive acquisition, non-ethical controversy, easy sampling and extraction, low immunogenicity, easy in vitro expansion, and have a stronger immunomodulatory function and stronger proliferation ability compared with other MSCs.

Given that the results of the published clinical studies so far are inconsistent and the outcome indicators of these clinical trials were not confirmed by the pathological results of kidney biopsy, investigators prompted to design a patient-blinded, randomized, placebo-controlled, parallel-design clinical trial (RCT) to test the safety and efficacy of MSC therapy for refractory lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old (including 18 and 65 years old, gender is not limited);
2. According to the revised criteria of ACR, the diagnosis of SLE was confirmed;
3. Diagnosed with LN (III, IV or III+V or IV+V) active lesions according to the 2016 revised ISN/RPS renal pathological classification criteria and unachieved a partial or complete response within 6-12 month of starting standard therapy.

   -

Exclusion Criteria:

1. Do not agree to sign the informed consent;
2. Pregnancy, lactation or do not agree to take effective contraceptive measures during the trial and within 12 months after the trial;
3. Kidney biopsy indicated chronic nephritis (extensive glomerular sclerosis, extensive fibrous crescent formation, extensive interstitial fibrosis, tubule atrophy);
4. In addition to SLE, patients with other autoimmune diseases (dermatomyositis/polymyositis, mixed connective tissue disease, scleroderma, rheumatoid arthritis, etc.);
5. Severe hepatic dysfunction (total bilirubin exceeding 14mg/L, AST or ALT exceeding 1.5 times the upper limit of normal) or estimated glomerular filtration rate (eGFR) ≤45ml/min per 1.73 m2;
6. Severe and uncontrollable cardiovascular disease, neurological disease, lung disease, endocrine or gastrointestinal disease;
7. Any substantial organ surgery performed within 12 weeks prior to screening is not tolerated by the test, or elective surgery is required during the study period;
8. A history of malignant tumors, including solid tumors and malignant hematological tumors (except resected or cured basal cell carcinoma of the skin, squamous cell carcinoma and cervical intraepithelial neoplasia);
9. A history of bone marrow, lung, liver, pancreas, or small intestine transplantation;
10. A current or recent (within 4 weeks prior to enrollment) history of serious active or recurrent bacterial, viral, fungal, parasitic or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, hepatitis B and C, HIV infection, shingles, but not tinea onychomycosis);
11. Had received live vaccine within 12 weeks prior to enrollment, or expected to require/receive live vaccine (other than shingles vaccine) during the study period;
12. Suffering from a serious mental illness (e.g. schizophrenia, bipolar personality disorder) that affects communication and decision-making;
13. Patients with severe allergies, who have a history of allergies to biological products, hypersensitivity reactions or other serious reactions;
14. Participate in other clinical trials within 30 days before enrollment.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Within 6-12 mo of starting therapy, but could take more than 12 mo
  * Number of participants with reduction in content of Protein creatinine ratio <0.5 g/g (50 mg/mmol) measured as the from of 24h-urine collection
  * Stabilization or improvement in kidney function (±10%-15% of baseline)
  * Within 6-12 month of starting therapy, but could take more than 12 month
Partial response rate | Within 6-12 mo of starting therapy
  * Number of participants with reduction in content of Protein creatinine ratio by at least 50% and to <3 g/g (300 mg/mmol) measured from a 24-h urine collection
  * Stabilization or improvement in kidney function (±10%-15% of baseline)
  * Within 6-12 mo of starting therapy
No kidney response rate | within 6-12 mo of starting therapy
  • Number of participants with failure to achieve a partial or complete response within 6-12 mo of starting therapy

SECONDARY OUTCOMES:
Number of participants with varying degrees of LN activity according to SLEDAI 2000 and BILAG 2004. | within 6-12 mo of starting therapy
  SLEDAI 2000: Systemic Lupus Erythematosus Disease Activity Index 2000 Totle score range from 0 to 105 Score 0-4 (Barely activity) Score 5-9 (Mild activity) Score 10-14 (Moderate activity) Score ≥15 (Severe activity)
  BILAG 2004: British Isles Lupus Assessment Group 2004 Index The system consists of 86 clinical indicators, and each system is distinguished by A, B, C, D, and E respectively.
  A, B, C, D, E is scored as follows: A=9, B=4, C=1, D=0, E=0. BILAG≥11 indicates active disease and BILAG<11 indicates stable for the disease.
Number of participants with the recurrence within 48 weeks after complete and partial remission. | within 6-12 mo of starting therapy
Number of participants with abnormal laboratory tests results for blood routine; blood biochemistry; urine routine; Immune indexes (ANA, Anti-dsDNA, C1q, C3, C4, etc.) and umor markers. | within 6-12 mo of starting therapy
Overall survival rate and survival rate without renal involvement. | within 6-12 mo of starting therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, Principal Investigator — Chinese PLA General Hospital